CLINICAL TRIAL: NCT01232803
Title: A Phase 1 Randomized, Double-Blinded, Placebo-Controlled Rectal Safety and Acceptability Study of Tenofovir 1% Gel
Brief Title: Rectal Safety and Acceptability Study of Tenofovir 1% Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MTN-007; 5U01AI068633-05 (NIH)
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Rectal Microbicides
Keywords: Rectal Microbicides; Tenofovir; Rectal use; Rectal mucosal damage
MeSH Terms: interventions — Tenofovir; Gels

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2% N-9 gel (Active Comparator): Rectal application of 2% N-9 gel
  Interventions: Drug: 2% N-9 gel
- HEC placebo gel (Placebo Comparator): Rectal application of HEC placebo gel
  Interventions: Drug: HEC Placebo gel
- no-treatment arm (No Intervention): no intervention
- Tenofovir 1% gel (Experimental): rectal application of Tenofovir 1% gel
  Interventions: Drug: Tenofovir 1% gel

INTERVENTIONS:
Drug: Tenofovir 1% gel — Entire contents of an applicator will be inserted rectally, for a total of 8 doses.
  Arms: Tenofovir 1% gel
Drug: 2% N-9 gel — Entire contents of an applicator will be inserted rectally, for a total of 8 doses.
  Arms: 2% N-9 gel
Drug: HEC Placebo gel — Entire contents of an applicator will be inserted rectally, for a total of 8 doses.
  Arms: HEC placebo gel

SUMMARY:
MTN-007 is a Phase 1, randomized, blinded, placebo-controlled safety and acceptability study of vaginally formulated tenofovir 1% gel (a reduced-glycerin formulation), when applied rectally. The primary objective of this study is to assess the safety of vaginally formulated tenofovir 1% gel when applied rectally.

After completing screening and baseline evaluation, eligible participants will be randomized to receive tenofovir 1% gel, 2% nonoxynol-9 gel (N-9) or placebo gel. The study will also include a no treatment arm. There will be 15 participants in each arm.

Participants will return to the clinic, where they will self-administer a single dose of the study gel under observation. Within approximately 30 minutes, lavage, stool, and rectal biopsy specimens will be obtained. After a one-week recovery period, participants will return to the clinic for assessment. If no significant adverse events (AEs) are reported they will begin to self-administer once-daily outpatient doses of the study gel for 7 days. Participants will return to clinic for evaluation and specimen collection after completion of 7 days of daily dosing.

DETAILED DESCRIPTION:
MTN-007 is a Phase 1, randomized, blinded, placebo-controlled safety and acceptability study of vaginally formulated tenofovir 1% gel (a reduced-glycerin formulation), when applied rectally. The primary objective of this study is to assess the safety of vaginally formulated tenofovir 1% gel when applied rectally. This study will also determine whether rectal use of tenofovir 1% gel is associated with rectal mucosal damage using a broad range of immunological safety biomarkers, utilizing N-9 as a positive control, as rectal application of N-9 is known to cause mild but transient mucosal damage. Other secondary objectives include evaluations of the acceptability of rectal administration of tenofovir 1% gel as well as the safety of hydroxyethylcellulose (HEC) placebo gel when applied rectally.

Participants will be randomized to receive a single dose of tenofovir 1% gel, 2% N-9 gel or a placebo gel that is applied by a clinician at the study site. The study will also include a no treatment arm. There will be 15 participants in each arm. Participants will return to the clinic, where they will self-administer a single dose of the study gel under observation. Within approximately 30 minutes, lavage, stool, and rectal biopsy specimens will be obtained. After a one-week recovery period, participants will return to the clinic for assessment. If no significant adverse events (AEs) are reported they will begin to self-administer once-daily outpatient doses of the study gel for 7 days. Participants will return to the clinic for evaluation and specimen collection after completion of 7 days of daily dosing.

Receptive anal intercourse is common among men who have sex with men and there is increasing evidence that heterosexual women in the developed and developing world also practice anal sex. It can therefore be anticipated that once vaginal microbicides are licensed, they will be used in both the vaginal and rectal compartments. As a consequence, there is a need to evaluate both the rectal and vaginal safety profile of candidate microbicides. The Rectal Microbicide Program clinical protocols have therefore been developed to assess the safety and pharmacology of tenofovir 1% gel when used rectally in men and women as well as address critical questions regarding rectal microbicides through exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ Age of 18 at screening, verified per site SOP
2. Willing and able to provide written informed consent for screening and enrollment
3. HIV-1 uninfected at screening
4. Willing and able to communicate in English
5. Willing and able to provide adequate locator information, as defined in site SOP
6. Availability to return for all study visits, barring unforeseen circumstances
7. Per participant report at screening, a history of consensual receptive anal intercourse (RAI) at least once in the prior year (Required to assure that participants have a context for the acceptability assessments).
8. Willing to abstain from insertion of anything rectally, including sex toys, other than the study gel for the duration of study participation
9. Willing to abstain from RAI for the duration of study participation
10. Must agree to use study provided condoms for the duration of the study for vaginal and insertive anal intercourse
11. Must be in general good health
12. At Screening and Enrollment, must agree not to participate in other research studies involving drugs, medical devices, or genital products for the duration of study participation (until all follow-up visits are completed) In addition to the criteria listed above, female participants must meet the following criteria:
13. Postmenopausal or using (or willing to use) an acceptable form of contraception (e.g., barrier method, intrauterine device (IUD), hormonal contraception, surgical sterilization, or vasectomization of male partner). If the female participant has female partners only, the method of contraception will be noted as a barrier method in the study documentation.

Exclusion Criteria:

1. Abnormalities of the colorectal mucosa, or significant colorectal symptom(s), which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition
2. At screening: participant-reported symptoms, and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current Centers for Disease Control (CDC) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic bacterial vaginosis, symptomatic vaginal candidiasis, other vaginitis, trichomoniasis, Chlamydia (CT), gonorrhea (GC), syphilis, active herpes simplex virus (HSV) lesions, chancroid, pelvic inflammatory disease, genital sores or ulcers, cervicitis, or symptomatic genital warts requiring treatment. Note that an HSV-1 or HSV-2 seropositive diagnosis with no active lesions is allowed, since treatment is not required Note: In cases of non-anorectal GC/CT identified at screening, one re-screening 2 months after screening visit will be allowed
3. Anorectal sexually transmitted infections (STI) within six months prior to the Screening Visit
4. At screening:

   Positive for hepatitis B surface antigen Hemoglobin < 10.0 g/dL Platelet count less than 100,000/mm3 White blood cell count < 2,000 cells/mm3 or > 15,000 cells/mm3 For females: calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min (140- age in years) x (weight in kg) x (0.85 for female)/72 x (serum creatinine in mg/dL) For males: calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min = (140 - age in years) x (weight in kg) x (1 for male)/72 x (serum creatinine in mg/dL) Serum creatinine > 1.3× the site laboratory upper limit of normal (ULN) Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5× the site laboratory ULN

   +1 glucose or +1 protein on urinalysis (UA) History of bleeding problems
5. History of significant gastrointestinal bleeding in the opinion of the investigator
6. Allergy to methylparaben, propylparaben, sorbic acid, and components of N-9
7. Known HIV-infected partners
8. By participant report at enrollment, history of excessive daily alcohol use (as defined by the CDC as heavy drinking consisting of an average consumption of more than 2 drinks per day for men, and more than 1 drink per day for women), frequent binge drinking or illicit drug use that includes any injection drugs, methamphetamines (crystal meth), heroin, or cocaine including crack cocaine, within the past 12 months
9. Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications during the period of study participation: Heparin, including Lovenox® Warfarin Plavix® (clopidogrel bisulfate) Rectally administered medications (including over-the-counter products) Aspirin Non-steroidal anti-inflammatory drugs (NSAIDS) Any other drugs that are associated with increased likelihood of bleeding following mucosal biopsy
10. By participant report at screening, use of post-exposure prophylaxis for HIV exposure, systemic immunomodulatory medications, rectally administered medications, rectally administered products (including condoms) containing N-9, or any investigational products within the 4 weeks prior to the Enrollment/Baseline Evaluation Visit and throughout study participation
11. History of recurrent urticaria
12. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease In addition to the criteria listed above, female participants will be excluded if they meet any of the following criteria:
13. Pregnant at the Enrollment/Baseline Visit
14. Breastfeeding at screening or intend to breastfeed during study participation per participant report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of tenofovir 1% gel when applied rectally | Duration of Study
  Grade 2 or higher AEs as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009) and/or Addenda 1 and 3 (Female Genital and Rectal Grading Tables for Use in Microbicide Studies)

SECONDARY OUTCOMES:
To evaluate the acceptability of tenofovir 1% gel when applied rectally | Duration of Study
  The proportion of participants who at their Final Clinic Visit report via the acceptability questionnaire that they would be very likely to use the candidate microbicide during receptive anal intercourse
To evaluate the safety of the placebo gel when applied rectally | Duration of Study
  Grade 2 or higher adverse events in the placebo gel arm, as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August MTN-007, Version 2.0 xii August 13, 2010 2009) and/or Addenda 1 and 3 (Female Genital and Rectal Grading Tables for Use in Microbicide Studies)
To determine whether use of tenofovir 1% gel is associated with rectal mucosal damage | Duration of Study
  Changes in the following parameters:
  * Epithelial sloughing
  * Intestinal histopathology
  * Intestinal mucosal mononuclear cell phenotype
  * Intestinal mucosal cytokine messenger RNA (mRNA)
  * Intestinal mucosal gene expression arrays
  * Cytokine profile in rectal secretions
  * Fecal calprotectin
  * Microflora
To determine whether use of 2% nonoxynol-9 gel (Gynol-II®) is associated with rectal mucosal damage | Duration of Study
  Changes in the following parameters:
  * Epithelial sloughing
  * Intestinal histopathology
  * Intestinal mucosal mononuclear cell phenotype
  * Intestinal mucosal cytokine messenger RNA (mRNA)
  * Intestinal mucosal gene expression arrays
  * Cytokine profile in rectal secretions
  * Fecal calprotectin
  * Microflora

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Fenway Institute, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] McGowan I, Hoesley C, Cranston RD, Andrew P, Janocko L, Dai JY, Carballo-Dieguez A, Ayudhya RK, Piper J, Hladik F, Mayer K. A phase 1 randomized, double blind, placebo controlled rectal safety and acceptability study of tenofovir 1% gel (MTN-007). PLoS One. 2013;8(4):e60147. doi: 10.1371/journal.pone.0060147. Epub 2013 Apr 3. PMID 23573238
- [Result] Leu CS, Mabragana M, Giguere R, Dolezal C, Carballo-Dieguez A, McGowan I. Use of a novel technology to track adherence to product use in a microbicide trial of short duration (MTN-007). AIDS Behav. 2013 Nov;17(9):3101-7. doi: 10.1007/s10461-013-0549-2. PMID 23842718
- [Result] Hladik F, Burgener A, Ballweber L, Gottardo R, Vojtech L, Fourati S, Dai JY, Cameron MJ, Strobl J, Hughes SM, Hoesley C, Andrew P, Johnson S, Piper J, Friend DR, Ball TB, Cranston RD, Mayer KH, McElrath MJ, McGowan I. Mucosal effects of tenofovir 1% gel. Elife. 2015 Feb 3;4:e04525. doi: 10.7554/eLife.04525. PMID 25647729